CLINICAL TRIAL: NCT02152501
Title: Exercise and Weight Control: A Search for Biological and Neurobehavioral Compensatory Mechanisms That Defend Against Exercise-Induced Negative Energy Balance
Brief Title: Exercise and Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC028
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obese
Keywords: obese; overweight; exercise; energy expenditure differences; relative reinforcing values (RRV); food; physical activity; biological; neurobehavioral; behavioral
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Energy Expenditure 300 kcal/day (Experimental): Subjects will be randomly assigned to this group and will exercise energy expenditure of 300 kcal/day.
  Interventions: Other: Exercise Energy Expenditure 300 kcal/day
- Exercise Energy Expenditure 600 kcal/day (Experimental): Subjects will be randomly assigned to this group and will exercise energy expenditure of 600 kcal/day.
  Interventions: Other: Exercise Energy Expenditure 600 kcal/day

INTERVENTIONS:
Other: Exercise Energy Expenditure 300 kcal/day
  Arms: Exercise Energy Expenditure 300 kcal/day
Other: Exercise Energy Expenditure 600 kcal/day
  Arms: Exercise Energy Expenditure 600 kcal/day

SUMMARY:
The purpose of this study is to research the effects of exercise on calories eaten and expended. The investigator expects to find out whether subjects change their eating and activity behaviors when starting an exercise program.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old
* BMI of 25.0 - 35 kg/m2
* willing to consent to study conditions
* not taking medications that affects energy expenditure or eating
* not using tobacco or nicotine products
* no food allergies or limitations to eating certain food that would prohibit them from eating the study foods
* not be dieting to lose weight
* no major health problems
* cannot have known cardiovascular, pulmonary or metabolic disease
* cannot be regularly exercising in an aerobic manner more than twice per week
* must have a liking of at least 5 out of 10 for 75% of the study foods

Exclusion Criteria:

* < 18 or > 40 years old
* BMI < 25 or >35 kg/m2
* currently pregnant or trying to become pregnant, or lactating
* currently using tobacco or nicotine
* taking medication that affects energy expenditure or eating
* food allergies to foods used in the study
* regularly exercising in an aerobic manner more than twice per week
* major health problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Negative Energy Balance as assessed by changes in adipose tissue | End Training (weeks 10-12)
  Whether participants were able to maintain a negative energy balance will be assessed by pre-post changes in stored adipose tissue, as assessed by a dual-energy x-ray absorptiometry scan (DEXA).

SECONDARY OUTCOMES:
Change in relative reinforcing value (RRV) of food | Pre-intervention (week 0) and End Training (weeks 10-12)
  RRV of food will be assessed by evaluating the number of responses (mouse button presses) a participant is willing to complete to gain access to food or an alternative sedentary activity.
Average daily calories consumed as assessed by dietary recall | Pre-intervention (week 0) and End Training (weeks 10-12)
  On two weekdays and one weekend day, participants will fill out the Automated Self-Administered 24-Hour Dietary Recall (ASA24) to estimate dietary intake (total energy, grams carbohydrates, fat, protein, alcohol).
Pre-post intervention changes in Ghrelin plasma levels | Pre-intervention (week 0) and End Training (weeks 10-12)
  Participants will provide a fasting blood sample collected in ethylenediaminetetraacetic acid (EDTA)-coated and serum tubes. Changes in acylated Ghrelin will be measured via enzyme-linked immunosorbent assay (ELISA).
Pre-post intervention changes in glucagon-like peptide 1 (GLP-1) plasma levels | Pre-intervention (week 0) and End Training (weeks 10-12)
  Participants will provide a fasting blood sample collected in EDTA-coated and serum tubes. Changes in GLP-1 concentrations will be measured via ELISA.
Pre-post intervention changes in Ghrelin concentrations | Pre-intervention (week 0) and End Training (weeks 10-12)
  Participants will provide a fasting blood sample collected in EDTA-coated and serum tubes. Changes in Ghrelin concentrations will be measured via ELISA.
Pre-post intervention changes in irisin concentrations | Pre-intervention (week 0) and End Training (weeks 10-12)
  Participants will provide a fasting blood sample collected in EDTA-coated and serum tubes. Changes in irisin concentrations will be measured via ELISA.
Pre-post intervention changes in myostatin plasma levels | Pre-intervention (week 0) and End Training (weeks 10-12)
  Participants will provide a fasting blood sample collected in EDTA-coated and serum tubes. Changes in myostatin levels will be measured via ELISA.
Change in relative reinforcing value (RRV) of physical activity | Pre-intervention (week 0) and End Training (weeks 10-12)
  RRV of physical activity will be assessed by evaluating the number of responses (mouse button presses) a subject is willing to complete to gain access to physical activity or a sedentary alternative.
Change in minutes of sedentary behavior, as assessed by activity tracker | Pre-intervention (week 0) and End Training (weeks 10-12)
  Minutes of sedentary behavior (non-exercise activity) will be assessed by having participants wear an Actigraph accelerometer for 7 days (minimum 10 hours per day) on the right hip.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA GFHNRC
Locations (1):
- USDA Grand Forks Human Nutrition Reserach Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No